CLINICAL TRIAL: NCT04823884
Title: Short-term Results After Minimally Invasive Chevron Osteotomy for Hallux Valgus Correction in Comparison to the Open Technique
Brief Title: Short-term Results After Minimally Invasive Chevron Osteotomy for Hallux Valgus Correction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr.Gerhard Kaufmann (Other)
Responsible Party: Sponsor-Investigator, Dr.Gerhard Kaufmann, Gerhard Kaufmann MD, Clinical Professor, OFZ Innsbruck
Organization: OFZ Innsbruck (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/1000
Record Dates: First submitted 2021-03-14; First posted 2021-04-01 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Hallux Valgus; Minimally Invasive Surgical Procedures
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: after completion of data collection personal data is anonymized. Outcomes assessor adds up the scores without knowing the type of surgery. The principal investigator as well as the statistical investigator do receive the completed anonymized excel file for doing the statistical analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open distal chevron osteotomy (Active Comparator): Hallux valgus correction is provided by using the traditional open distal v-shaped chevron osteotomy.
  Interventions: Procedure: open distal chevron osteotomy
- minimally invasive distal chevron osteotomy (Active Comparator): Hallux valgus correction is provided by using a minimally invasive distal v-shaped chevron osteotomy.
  Interventions: Procedure: minimally invasive distal chevron osteotomy

INTERVENTIONS:
Procedure: open distal chevron osteotomy — Through a 4-cm-long dorsomedial skin incision the V-shaped osteotomy with the apex 1-2 mm superior to the center of the metatarsal head is performed. The angle of the chevron is 60° to 90°. The direction of the osteotomy is angled toward the center of the third metatarsal head. After shifting the metatarsal head laterally, fixation is achieved by usage of one cannulated screw (3.0 mm or 2.5mm). Prominent bone ridges are resected with a saw. A distal soft tissue procedure is performed in every case through the same skin incision. The adductor hallucis tendon is detached from its insertion at the phalangeal bone and from the lateral border of the fibular sesamoid. The transverse intermetatarsal ligament is released and a T-shaped capsulotomy is performed to allow reposition of the sesamoids. Sesamoid position is controlled by sight. After closing of the medial capsula skin is closed with nylon sutures.
  Other Names: austin osteotomy
  Arms: open distal chevron osteotomy
Procedure: minimally invasive distal chevron osteotomy — The osteotomy is performed percutaneously through a dorsomedial incision of 3-5 mm. An electric motor-driven machine used for the osteotomy. To prevent overheating the reamer is frequently rinsed with sterile saline. The medial eminence is excised and the V-shaped osteotomy is performed. The apex of the osteotomy is identified by fluoroscopy and centered 1-2 mm superior to the center of the metatarsal head. The angle of the osteotomy amounts to 60-90 degrees as well. Bone debris is washed out with sterile saline. A lateral soft-tissue release is undertaken through a separate lateral incision of 3-5 mm. The distal fragment is shifted laterally and fixed with a canulated screw of 3.5mm. Residual bone ridges are reamed. Position of the metatarsal head and the K-wire is controlled by fluoroscopy. The skin is closed with a nylon sutures.
  Arms: minimally invasive distal chevron osteotomy

SUMMARY:
By means of clinical satisfaction and clinical scores comparison of an open to a minimally invasive distal chevron osteotomy for correction of a hallux valgus deformity is performed.

DETAILED DESCRIPTION:
The aim of this study is to evaluate shortterm clinical outcome after a minimally invasive chevron osteotomy technique for correction of hallux valgus deformity in comparison to the open distal chevron technique. Patients undergoing a distal chevron osteotomy for correction of a hallux valgus deformity are assigned to one of the two groups. Survey is taken preoperatively, after 2, 4, 6 and 12 weeks postoperatively. Assessment of the clinical outcome measures in terms of the range of motion (ROM), Visual Analogue Scores (VAS) of pain, the American Orthopaedic Foot and Ankle Society (AOFAS) forefoot Score and a patient satisfaction score and a Life Quality score (SF 12) as well as the evaluation of the Charlson Comorbidity score is performed. It is hypothesized, that clinical outcome with the minimally invasive distal chevron osteotomy is superior to the open technique.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing hallux valgus correction by means of a distal chevron osteotomy

Exclusion Criteria:

* surgery on the lesser rays of the same foot
* mental illness with impossibility to follow the postoperative protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical outcome after correction of hallux valgus deformity within the first three months after surgery: a comparison of the minimally invasive versus the open distal chevron osteotomy technique . | Change of the scores from preoperative to postoperative at 2 weeks, 4 weeks, 6 and 12 weeks is measured
  Clinical outcome is assessed for both techniques with a clinical score to specific time points.
  AOFAS Hallux etmatarsophalangeal -interphalangeal Scale [maximum 100 points, minimum 0 points - higher scores mean better outcome]
Clinical outcome after correction of hallux valgus deformity within the first three months after surgery: a comparison of the minimally invasive versus the open distal chevron osteotomy technique . | Change of the scores from preoperative to postoperative at 2 weeks, 4 weeks, 6 and 12 weeks is measured
  Clinical outcome is assessed for both techniques with a clinical score to specific time points.
  Maryland Foot Score [maximum 100 points, minimum 0 points - higher scores mean better outcome]
Clinical outcome after correction of hallux valgus deformity within the first three months after surgery: a comparison of the minimally invasive versus the open distal chevron osteotomy technique . | Change of the score from preoperative to postoperative at 2 weeks, 4 weeks, 6 and 12 weeks is measured
  Clinical outcome is assessed for both techniques with clinical a score to specific time points.
  JSSF Hallux metatarsophalangeal -interphalangeal Scale [maximum 100 points, minimum 0 points - higher scores means better outcome]
Clinical outcome after correction of hallux valgus deformity within the first three months after surgery: a comparison of the minimally invasive versus the open distal chevron osteotomy technique . | Change of the SF 12 score from preoperative to postoperative at 2 weeks, 4 weeks, 6 and 12 weeks is measured
  Clinical general situation is assessed for both techniques to specific time points by using the SF12 Life Quality Score [maximum 47 points, minimum 0 points - higher scores mean better clinical situation]
Clinical outcome after correction of hallux valgus deformity within the first three months after surgery: a comparison of the minimally invasive versus the open distal chevron osteotomy technique . | Change of the VAS from preoperative to postoperative at 2 weeks, 4 weeks, 6 and 12 weeks is measured
  Clinical outcome and therefore the pain level is assessed for both techniques to specific time points by using the Visual Analogue Score for pain [0-10])
Clinical outcome after correction of hallux valgus deformity within the first three months after surgery: a comparison of the minimally invasive versus the open distal chevron osteotomy technique . | Change of the range of motion and therefore the clinical outcome from preoperative to postoperative at 2 weeks, 4 weeks, 6 and 12 weeks is measured
  Clinical outcome is assessed for both techniques to specific time points by assessing the Range of motion (normal range 70-0-45 degrees)
Clinical outcome after correction of hallux valgus deformity within the first three months after surgery: a comparison of the minimally invasive versus the open distal chevron osteotomy technique . | Change of the foot circumference at the level of surgery from preoperative to postoperative at 2 weeks, 4 weeks, 6 and 12 weeks is measured
  Clinical outcome and therefore changes of the foot circumference at the level of surgery is assessed for both techniques to specific time points by measuring the foot circumference at the level of surgery (measurement in centimeter).

OTHER OUTCOMES:
Clinical outcome after correction of hallux valgus deformity within the first three months after surgery: a comparison of the minimally invasive versus the open distal chevron osteotomy technique . | This score is used to compare the clinical fitness of both cohorts preoperatively.
  Clinical fitness of our cohort is assessed by means of the Charlson Comorbidity Index [maximum 37 points, minimum 0 points - lower scores mean clinical situation] preoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Priv-Doz. Dr. Gerhard Kaufmann, Innsbruck, Tyrol, Austria